CLINICAL TRIAL: NCT06405438
Title: Comparison of the Efficacy of Peloid Therapy and Paraffin Treatment in Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; median neuropathy; median nerve; peloid therapy; mud therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peloid therapy group: Patients in this group have already received peloid therapy for their carpal tunnel syndrome. Peloid therapy involves the application of natural mud, typically rich in minerals, to the affected area. The sessions will also last approximately 20-30 minutes per day, administered consecutively for 5 days a week, totaling 10 sessions for 2 weeks.
  Interventions: Other: No intervention
- Paraffin treatment group: In this group, patients have already received paraffin treatment for their carpal tunnel syndrome. Paraffin treatment involves immersing the affected hand or hands in a mixture of heated paraffin wax. The sessions will last approximately 20-30 minutes per day, 5 days a week, for a total of 15 sessions for 3 weeks.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
This study compares the effectiveness of peloid therapy and paraffin treatment in carpal tunnel syndrome. Patients who have already received 2 weeks of peloid therapy or 15 sessions of paraffin treatment will be assessed. Pain and symptom severity are assessed using the Visual Analog Scale (VAS) and Boston Carpal Tunnel Syndrome Questionnaire (BCTQ). Electrophysiological examinations will also be conducted at the same time points: baseline, 4 weeks post-treatment, and a 12-week follow-up.

DETAILED DESCRIPTION:
Our study will include 60 patients aged 18-65 who visited the outpatient clinics of Beylikdüzü State Hospital between January 1, 2024, and September 1, 2024, and were diagnosed with mild to moderate carpal tunnel syndrome based on electrophysiological examinations. These patients received either peloid or paraffin treatment. Patients with symptoms persisting for a minimum of 3 months will be included in the study. In this study, pain levels will be evaluated using the Visual Analog Scale (VAS), and the type and severity of symptoms will be assessed with the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ). At our hospital, the standard paraffin treatment consists of 15 sessions, administered 5 days per week, while the peloid therapy consists of 10 sessions, also administered 5 days per week. The VAS, BCTQ scores, and electrophysiological evaluations of the patients will be assessed at the 4th and 12th weeks post-treatment. Electrophysiological parameters including median nerve distal motor latency (MMNDL), median nerve distal sensory latency (MNSDL), sensory nerve conduction velocity (SNCV), compound muscle action potential (CMAP), and sensory nerve action potential (SNAP) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years old.
* Patients diagnosed with mild to moderate carpal tunnel syndrome based on electrophysiological evaluations.
* Patients experiencing symptoms for a minimum of 3 months.

Exclusion Criteria:

* Patients diagnosed with neuropathic conditions such as polyneuropathy, brachial plexopathy, or thoracic outlet syndrome.
* Patients with a history of previous injections or surgery for carpal tunnel syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild and moderate carpal tunnel syndrome
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | 0 day, 4th week and 12th week
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) consists of two parts: the Symptom Severity Scale (SSS) and the Functional Status Scale (FSS). Both parts are scored on a 5-point Likert scale, with higher scores indicating worse symptoms or functional impairment.The highest possible total score for the Symptom Severity Scale is 55, which reflects the most severe symptoms.The highest possible total score for the Functional Status Scale is 40, indicating the greatest functional impairment.The minimum total score is 19 (indicating minimal or no symptoms and functional limitations).
  The maximum total score is 95 (indicating the most severe symptoms and functional limitations).
  As the total score increases, the severity of symptoms and functional limitations worsens, meaning higher scores reflect worse outcomes.

SECONDARY OUTCOMES:
Visual Analogue Scale | 0 day, 4th week and 12th week
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain.
  The Visual Analog Scale (VAS) is a tool used to measure pain intensity. It is typically represented as a 10 cm or 100 mm line, where the patient marks their pain level.
  The minimum score is 0, which indicates no pain. The maximum score is 100, indicating the worst possible pain. As the score increases, the severity of pain worsens. In this scale, higher scores reflect more intense pain levels. The Visual Analog Scale (VAS) ranges from 0 to 100 where higher scores reflect greater pain intensity.
Median nerve distal motor latency | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Median nerve distal sensory latency | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Sensory nerve conduction velocity | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Motor nerve conduction velocity | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Sensory nerve action potential amplitude | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Motor nerve action potential amplitude | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Şirin Ahısha, MD, Principal Investigator — Beylikdüzü State Hospital
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No